CLINICAL TRIAL: NCT06073886
Title: Personalized Circuit-Based Frontoamygdala Neuromodulation for Persistent Post-Concussive Symptoms
Brief Title: Personalized Brain Stimulation to Treat Chronic Concussive Symptoms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kevin Charles Bickart, MD, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP210602
Record Dates: First submitted 2023-04-20; First posted 2023-10-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Post-Concussion Syndrome; Concussion, Brain; Mild Traumatic Brain Injury; Head Injury; Headache; Dizziness; Cognitive Symptom; Dysautonomia; Anxiety; Irritability; Syndrome; Depression; Post-traumatic Stress Disorder
Keywords: Transcranial Magnetic Stimulation; Magnetic Resonance Imaging; Functional MRI; Personalized neuromodulation; Amygdala; Prefrontal Cortex
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion; Craniocerebral Trauma; Headache; Dizziness; Neurobehavioral Manifestations; Autonomic Nervous System Diseases; Anxiety Disorders; Syndrome; Depression; Stress Disorders, Post-Traumatic | interventions — Implosive Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Active continuous theta-burst stimulation (cTBS) plus exposure (Experimental): 10 days of active, continuous theta-burst stimulation (cTBS) will be delivered to a personalized region of the ventromedial prefrontal cortex (vmPFC) based on baseline brain circuit mapping for each individual participant.
  Interventions: Device: Active cTBS; Behavioral: Imaginal exposure
- Inactive/Sham continuous theta-burst stimulation (cTBS) plus exposure (Sham Comparator): 10 days of inactive, or sham, continuous theta-burst stimulation (cTBS) will be delivered to a personalized region of the ventromedial prefrontal cortex (vmPFC) based on baseline brain circuit mapping for each individual participant.
  Interventions: Device: Inactive/Sham cTBS; Behavioral: Imaginal exposure
- Active Comparator continuous theta-burst stimulation (cTBS) plus exposure (Active Comparator): 10 days of active, continuous theta-burst stimulation (cTBS) will be delivered to a personalized region of the ventromedial prefrontal cortex (vmPFC) based on baseline brain circuit mapping for each individual participant.
  Interventions: Device: Active cTBS; Behavioral: Imaginal exposure

INTERVENTIONS:
Device: Active cTBS — 600 active cTBS pulses will be delivered continuously (3 pulses at 50 hertz (Hz), repeated at 5 Hz, 15 pulses/sec, continuously for 40 seconds) twice/day for 1,200 pulses/day. The MagVenture MagPro active/sham system will be used to enable double blinding by universal serial bus (USB) key in which a current will be delivered through surface electrodes on the skin beneath the coil to mimic the sensory experience of cTBS for active and sham groups.
  Arms: Active Comparator continuous theta-burst stimulation (cTBS) plus exposure; Active continuous theta-burst stimulation (cTBS) plus exposure
Device: Inactive/Sham cTBS — 600 inactive, or sham, cTBS pulses will be delivered continuously (3 pulses at 50 hertz (Hz), repeated at 5 Hz, 15 pulses/sec, continuously for 40 seconds) twice/day for 1,200 pulses/day. The MagVenture MagPro active/sham system will be used to enable double blinding by universal serial bus (USB) key in which a current will be delivered through surface electrodes on the skin beneath the coil to mimic the sensory experience of cTBS for active and sham groups.
  Arms: Inactive/Sham continuous theta-burst stimulation (cTBS) plus exposure
Behavioral: Imaginal exposure — Personalized recordings about participants' descriptions of triggering or neutral stimuli or activities

SUMMARY:
The goal of this study is to investigate a new treatment for chronic symptoms after concussion or mild traumatic brain injury in people aged 18-65 years old. Chronic symptoms could include dizziness, headache, fatigue, brain fog, memory difficulty, sleep disruption, irritability, or anxiety that occurred or worsened after the injury. These symptoms can interfere with daily functioning, causing difficulty returning to physical activity, work, or school. Previous concussion therapies have not been personalized nor involved direct treatments to the brain itself. The treatment being tested in the present study is a noninvasive, personalized form of brain stimulation, called transcranial magnetic stimulation (TMS).

The investigators intend to answer the questions:

1. Does personalized TMS improve brain connectivity after concussion?
2. Does personalized TMS improve avoidance behaviors and chronic concussive symptoms?
3. Do the improvements last up to 2 months post-treatment?
4. Are there predictors of treatment response, or who might respond the best?

Participants will undergo 14 total visits to University of California Los Angeles (UCLA):

1. One for the baseline symptom assessments and magnetic resonance imaging (MRI)
2. Ten for TMS administration
3. Three for post-treatment symptom assessments and MRIs

Participants will have a 66% chance of being assigned to an active TMS group and 33% chance of being assigned to a sham, or inactive, TMS group. The difference is that the active TMS is more likely to cause functional changes in the brain than the inactive TMS.

DETAILED DESCRIPTION:
The overall objective of the proposed project is to apply a well-studied and safe form of brain modulation to patients with chronic symptoms after concussion. These patients represent a vulnerable population in need of brain-targeted and personalized therapies. Chronic concussive symptoms can include emotional, physical, and cognitive problems, such as depression, anxiety, headache, dizziness, sensory sensitivities, and difficulties with memory and attention. These symptoms are costly and relatively common, representing a public health concern, yet there are no standard therapies. This is in part due to a limited understanding of the underlying cause of these symptoms.

Most concussions do not cause a visible injury to the brain based on clinical-grade brain imaging. Using research-grade brain imaging however, the investigators have identified an overactive brain circuit in patients who have more chronic symptoms after concussion and more severe forms of traumatic brain injury. Interestingly, this brain circuit connects the frontal lobe of the brain to a deep structure in the brain, called the amygdala, which is important for generating and regulating emotions. The investigators' finding suggests that this brain circuit may be involved in chronic concussive symptoms. This is promising because the frontal lobe can be targeted with noninvasive brain modulation treatment. In fact, these preliminary findings show that inhibiting the frontal lobe at the midline, over the forehead, can decrease the activity of this brain circuit.

Whereas these preliminary findings are promising, this target location and modulation technique have not been studied in patients with concussion. Here, the investigators propose leveraging this prior work to apply the same brain modulation approach to patients with chronic symptoms after concussion. The investigators will also advance this approach to personalize the brain modulation and optimize chances of modulating the intended brain circuit by mapping each individual's brain circuits prior to treatment. The study will be conducted in patients between 18 and 65 years old who have had a mild traumatic brain injury, including concussion, and report a significant burden of symptoms up to 12 months after their injury.

Seventy-five participants will be randomly assigned to active modulation and sham modulation (or inactive in which the participant receives only a sensation of brain modulation without actual modulation) groups. The investigators hypothesize that active brain modulation, as compared to sham modulation, will cause a decrease in activity in the brain circuit that the investigators found to be abnormally overactive in their prior studies of patients with chronic concussive symptoms. Furthermore, the investigators hypothesize that this personalized approach to frontal brain modulation will cause an improvement in chronic concussive symptoms in the active modulation but not sham modulation group, and that the improvements would be greatest for participants who showed the greatest decrease in activity of the targeted brain circuit. Finally, the investigators will also have collected many other data points about each individual that would allow us to determine what individual characteristics make one more likely to respond to this type of treatment.

This would be the first study to use brain circuit mapping on an individual level to treat patients with chronic concussive symptoms. It would not only have implications in this patient population but also any population that suffers from emotion regulation problems, such as in mood and anxiety disorders. Based on the investigators' analyses of treatment response, the investigators may even be able to determine which people would be most likely to respond to this form of frontal lobe modulation prior to recommending the treatment, a key prerequisite for precision medicine. Importantly, the findings from this work would be directly relevant to military personnel because of their higher risk of incurring combined physical and psychological trauma in battle and the higher prevalence of combined post-traumatic stress disorder and chronic concussive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Mild traumatic brain injury (mTBI) defined in accord with the World Health Organization criteria in the last 12 months
* age 18-65 at the time of the mTBI
* high burden of post-concussive symptoms defined as a score >=20 on the Rivermead Post-Concussion Symptoms Questionnaire

Exclusion Criteria:

* objective neurologic deficits
* ongoing or prolonged (>3 months) post-concussive symptoms from a prior mTBI within 2 years of the index injury
* history of transcranial magnetic stimulation (TMS) therapy
* contraindications for TMS or magnetic resonance imaging (MRI) (e.g., metallic implant other than dental, pacemaker)
* severe mental, physical, or medical problems that would impede participation or pose a risk for the planned intervention (e.g., liver, kidney, or heart disease, uncontrolled diabetes or hypertension, malignancy, psychosis, previous seizure, pregnancy)
* active alcohol or illicit drug abuse
* inability to speak and read English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Central target engagement, modulation, and durability | Change from baseline across all subsequent time points until completion of the study, an average of 4 months
  Using resting-state functional magnetic resonance connectivity in the target frontoamygdala circuit
Peripheral target engagement, modulation, and durability | Change from baseline across all subsequent time points until completion of the study, an average of 4 months
  Using heart rate variability as measured by electrocardiogram
Persistent post-concussive symptoms modulation and durability | Change from baseline across all subsequent time points until completion of the study, an average of 4 months
  Using the Modified Rivermead Post Concussion Symptoms Questionnaire where higher scores are worse. Scores range from 0-64.
Fear avoidance modulation and durability | Change from baseline across all subsequent time points until completion of the study, an average of 4 months
  Using the Fear Avoidance Behavior Questionnaire for Traumatic Brain Injury where higher scores are worse. Scores range from 0-48.

SECONDARY OUTCOMES:
Nightly Sleep Score from Oura Ring | Change from baseline across all subsequent time points until completion of the study, an average of 4 months
  Using sleep quality metric, called Sleep Score, from the Oura Ring where higher scores are better, ranging from 0-100.
Daily heart rate variability | Change from baseline across all subsequent time points until completion of the study, an average of 4 months
  Using heart rate variability metric from the Oura Ring
Weekly avoidance behavior | Change from baseline across all subsequent time points until completion of the study, an average of 4 months
  Using a single item question "I avoid activities that might make my symptoms worse" where higher ratings are worse. Ratings range from 1-10.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Westwood, Los Angeles, California, United States

REFERENCES:
- [Background] Bickart KC, Olsen A, Dennis EL, Babikian T, Hoffman AN, Snyder A, Sheridan CA, Fischer JT, Giza CC, Choe MC, Asarnow RF. Frontoamygdala hyperconnectivity predicts affective dysregulation in adolescent moderate-severe TBI. Front Rehabil Sci. 2023 Jan 4;3:1064215. doi: 10.3389/fresc.2022.1064215. eCollection 2022. PMID 36684686